CLINICAL TRIAL: NCT02658578
Title: Peripheral Nerve Stimulation and Motor Training to Enhance Hand Function After Stroke
Brief Title: Peripheral Nerve Stimulation and Motor Training in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação Faculdade de Medicina (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Adriana Bastos Conforto, Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0546/2011; R01NS076348 (NIH)
Record Dates: First submitted 2015-12-29; First posted 2016-01-20 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2020-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active PNS (Active Comparator): Active PNS will be administered by 2 pairs of surface electrodes (cathode proximal). One pair will overly the median and ulnar nerves at the wrist, and the other pair will overly the radial nerve. Trains of electric stimulation will be delivered at 1 Hz by using isolation units connected to a square pulse stimulator.
  Interventions: Procedure: PNS
- Sham PNS (Placebo Comparator): In sham PNS, the median, ulnar and radial nerves will not be actively stimulated.
  Interventions: Procedure: PNS

INTERVENTIONS:
Procedure: PNS — Active PNS will be administered by 2 pairs of surface electrodes (cathode proximal). One pair will overly the median and ulnar nerves at the wrist, and the other pair will overly the radial nerve. Trains of electric stimulation will be delivered at 1 Hz by using isolation units connected to a square pulse stimulator. In sham PNS, the median, ulnar and radial nerves will not be actively stimulated.
  Other Names: Peripheral Nerve Stimulation

SUMMARY:
Cerebrovascular disease is a major cause of disability worldwide. The catastrophic burden of stroke is more dramatic in low- and middle- income countries, and the scarcity of evidence-based rehabilitation interventions represents a major challenge to global health care. Upper limb weakness is frequent after stroke, but there is no universally accepted treatment to effectively improve hand function in patients with moderate and severe motor impairment. These are the patients in deepest need of rehabilitative interventions. This project addresses this important issue, by testing effects of a novel approach. The investigators will non-invasively stimulate peripheral nerves in order to enhance effects of motor training aided by an electrical stimulation device in patients with moderate to severe hand weakness. Our hypothesis is that peripheral nerve stimulation will enhance effects of motor training in patients in the chronic stage after stroke.

DETAILED DESCRIPTION:
The objective of this protocol is to determine whether a neuromodulation intervention associated with functional electrical stimulation, when combined with task-specific training over several sessions, decreases upper limb motor disability, motor impairment, overall disability and improves quality of life compared to the sham intervention and functional electrical stimulation.

The interventions will consist of three sessions per week, over six weeks, of outpatient functional electrical stimulation of the paretic wrist and task-specific training. In each session, either active peripheral nerve stimulation (PNS) or sham PNS will be applied. Before the first session, patients will be familiarized with the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age, 18 years or older;
* Ischemic or hemorrhagic stroke at least six months before, confirmed by computed tomography or magnetic resonance imaging;
* Moderate to severe motor impairment of an upper limb, defined as a score between 7 and 50 on the Fugl-Meyer Assessment of Sensorimotor Recovery after stroke, a scale with scores for upper limb ranging from 0 (no function) to 66 (normal function);
* Ability to provide written Informed Consent (patient or legal representative);
* Ability to comply with the schedule of interventions and evaluations in the protocol.

Exclusion Criteria:

* Lack of ability to voluntarily activate any active range of wrist extension;
* Anesthesia of the paretic hand;
* Severe spasticity at the paretic elbow, wrist, or fingers, defined as a score of >3 on the Modified Ashworth Spasticity Scale;
* Active joint deformity;
* Uncontrolled medical problems such as end-stage cancer or renal disease;
* Pregnancy;
* Seizures, if current use of drugs that may decrease seizure threshold such as tryciclic antidepressants;
* Pacemakers;
* Other neurological disorders such as Parkinson's disease;
* Psychiatric illness including severe depression;
* Aphasia or serious cognitive deficits that preclude comprehension of the experimental protocol or ability to provide consent;
* Treatment of upper limb spasticity with botulinum toxin within the past three months.
* Lesions that affect the cerebellum or cerebelar/vestibular pathways in the brainstem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Wolf Motor Function Test | 6 weeks
  The primary outcome will be evaluated before the intervention and 6 weeks after the beginning of the intervention.

SECONDARY OUTCOMES:
Motor Activity Log | 18 weeks
  This questionnaire will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Active range of motion of wrist extension in the paretic side | 18 weeks
  This physiological parameter will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Active range of motion of wrist flexion in the paretic side | 18 weeks
  This physiological parameter will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Grasp force in the paretic side | 18 weeks
  This physiological parameter will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Grip force in the paretic side | 18 weeks
  This physiological parameter will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Fugl-Meyer Assessment of Sensorimotor Recovery | 18 weeks
  This scale will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Barthel Index | 18 weeks
  This scale will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Stroke Impact Scale | 18 weeks
  This scale will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Beck Depression Inventory-short Form | 18 weeks
  This questionnaire will be evaluated before the intervention and 3, 6, 10 and 18 weeks after the beginning of the intervention.
Wolf Motor Function Test | 18 weeks
  This scale as a secondary outcome will be evaluated before the intervention and 3, 10 and 18 weeks after the beginning of the intervention.
Modified Ashworth Scale | 18 weeks
  This scale will be evaluated before the intervention and 3, 6, 10 and 18 weeks
Minimal Clinically Important Difference - Wolf Motor Function Test - time | 18 weeks
  This outcome will be evaluated at 6, 10 and 18 weeks
Minimal Clinically Important Difference - Wolf Motor Function Test - Functional Ability Scale | 18 weeks
  This outcome will be evaluated at 6, 10 and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Conforto, MD PhD, Principal Investigator — Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo/ Fundação Faculdade de Medicina
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo/Fundação Faculdade de Medicina, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Conforto AB, Machado AG, Ribeiro NHV, Plow EB, Liew SL, da Costa Leite C, Zavaliangos-Petropulu A, Menezes I, Dos Anjos SM, Luccas R, Peckham PH, Cohen LG. Repetitive Peripheral Sensory Stimulation as an Add-On Intervention for Upper Limb Rehabilitation in Stroke: A Randomized Trial. Neurorehabil Neural Repair. 2021 Dec;35(12):1059-1064. doi: 10.1177/15459683211046259. Epub 2021 Sep 29. PMID 34587830
- [Derived] Conforto AB, Machado AG, Menezes I, Ribeiro NHV, Luccas R, Pires DS, Leite CDC, Plow EB, Cohen LG. Treatment of Upper Limb Paresis With Repetitive Peripheral Nerve Sensory Stimulation and Motor Training: Study Protocol for a Randomized Controlled Trial. Front Neurol. 2020 Mar 25;11:196. doi: 10.3389/fneur.2020.00196. eCollection 2020. PMID 32269549